CLINICAL TRIAL: NCT06949189
Title: Nail Bed Repair With or Without Nail Bed Coverage: Randomized Clinical Trial
Brief Title: Nail Bed Repair With or Without Nail Bed Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patel Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Osheen Abbasi, Principal Investigator, Department of Plastic Surgery, Patel Hospital, Karachi, Patel Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH/IRB/2023/042
Record Dates: First submitted 2025-04-12; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Infection; Laceration Repair; Laceration Repair, Children; Nail Bed Injury
Keywords: nail bed repair; nail bed coverage; infection after nail bed repair; fingertip laceration; pediatric nail bed injury; randomized clinical trial
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nail bed coverage (Experimental): Following debridement and suturing of the nail bed, the fingernail will be replaced and secured with a figure-of-eight suture using Prolene. A low-adherent dressing will be applied. If the fingernail is unavailable (e.g., due to damage or loss), a substitute material (such as foil) will be chosen by the operating surgeon
  Interventions: Procedure: Nail Bed Repair with Nail Bed Coverage
- No Nail Bed Coverage (Active Comparator): Following debridement and suturing of the nail bed, the fingernail will be discarded. A low-adherent dressing will be applied without any covering of the nail bed
  Interventions: Procedure: Nail Bed Repair without Nail Bed Coverage

INTERVENTIONS:
Procedure: Nail Bed Repair with Nail Bed Coverage — Following debridement and suturing of the nail bed, the fingernail will be replaced and secured with a figure-of-eight suture using Prolene. A low-adherent dressing will be applied. If the fingernail is unavailable (e.g., due to damage or loss), a substitute material (such as foil) will be chosen by the operating surgeon
  Other Names: Nail Plate Repositioning; Nail Bed Coverage
  Arms: nail bed coverage
Procedure: Nail Bed Repair without Nail Bed Coverage — Following debridement and suturing of the nail bed, the fingernail will be discarded. A low-adherent dressing will be applied without any covering of the nail bed
  Other Names: No Nail Bed Coverage; Nail Plate Discarding
  Arms: No Nail Bed Coverage

SUMMARY:
A randomized clinical trial conducted at Patel hospital, Karachi, from March 2024 to February 2025, to evaluate infection in patients undergoing nailbed repair with and without nailbed coverage, with minimum follow up for one month post operative.

DETAILED DESCRIPTION:
Background:

The fingernail serves as a protective barrier for the dorsal fingertip while also enhancing its aesthetic appeal. Fingertip injuries account for approximately two-thirds of pediatric hand injuries, with nail bed injuries comprising 15% to 24% of these cases. In the United Kingdom, 96% of surgeons routinely remove the nail plate, repair the nail bed, and reposition the nail plate onto the nail bed. The rationale for repositioning includes protecting the repair, reducing infection risk, minimizing pain during dressing changes, and preventing adhesions by supporting the nail fold. When the autologous nail is unavailable, alternatives such as silver foil is used.

Objective:

This study aims to evaluate the risk of surgical site infection after nail bed repair with and without nail bed coverage.

Methods:

This is a two-arm randomized clinical trial enrolling 152 patients (76 in each group) over a 12-month period from March 2024 to February 2025. Patients undergoing nail bed repair will be randomized into two groups-one receiving nail bed coverage (repositioned nail or substitute) and the other without coverage. The primary outcome is the incidence of surgical site infection. Secondary outcomes include pain during dressing changes and cosmetic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all age groups and genders,
* Presented to the emergency or outpatient department within 48 hours of injury,
* Provided written informed consent (or had consent given by a parent/guardian in the case of minors),
* Injury to a single finger,
* Fractures that do not involve an open wound or require fixation.

Exclusion Criteria:

* Infected injuries,
* Underlying nail diseases,
* Pre-existing deformities in the injured or contralateral finger,
* Distal phalanx fractures requiring fixation,
* Amputations,
* Partial or complete loss of the nail bed requiring reconstruction,
* Multiple nail bed injuries,
* Known allergies to prescribed postoperative medications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
infection | 30 days
  Surgical site infection (SSI) was diagnosed according to CDC guidelines, requiring at least two of the following criteria within 30 days postoperatively:
  * Purulent discharge
  * Pain, with a numerical pain scale value of 7 or greater considered positive
  * Swelling
  * Erythema, defined as visible redness extending beyond the distal interphalangeal joint compared to the contralateral finger
  * Tenderness, characterized by pain upon touch

CONTACTS AND LOCATIONS:
Locations (1):
- Patel Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
patient confidentiality